CLINICAL TRIAL: NCT03918668
Title: Observational Study to Understand the Risk Factors Associated With Breast Cancer in Women With a Recent Diagnosis at the Community of Madrid
Brief Title: Study for the Knowledge of Risk Factors Associated With Breast Cancer in Women
Acronym: Mamanut
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI-2842
Record Dates: First submitted 2019-02-28; First posted 2019-04-17 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2019-02

CONDITIONS: Breast Neoplasm Female; Nutrition Related Cancer; Habits, Diet; Cancer, Breast
Keywords: breast neoplasm; cancer; risk factor; nutrition
MeSH Terms: conditions — Feeding Behavior; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Women with recent diagnosis of breast cancer — To evaluate dietary habits of a group of women with pre and post-surgical breast cancer

SUMMARY:
Breast cancer is the most frequent tumor in Western women. In Spain about 26,000 new breast cancers are diagnosed each year. This type of tumor is increasing worldwide with an increase in aggressive neoplasms in young women. There are some risk factors responsible for this global increase: lifestyle, diet and body weight especially in postmenopausal women.

Some cell mutations, especially in the BRCA1, BRCA2 and p53 genes, are associated with a very high risk of this type of cancer. Some authors have calculated the contribution of various modifiable risk factors to the global burden of breast cancer, and they concluded that 21% of all breast cancer deaths are attributable to alcohol consumption, overweight and obesity, and lack of physical activity. Nowadays, there aren't specific studies in the Community of Madrid designed to know the risk factors related to breast cancer.

For this reason, it is proposed to carry out an observational study that collects detailed information about dietary habits, genetic factors and life quality of a group of women with recent diagnosis in pre or post-surgical phase.

DETAILED DESCRIPTION:
1. Storage of biological sample at the Hospital.
2. Patient's breast pathology characteristics.
3. Study of concomitant pathologies.
4. Dietary study: "Frequency of Food Consumption" questionnaire referring to the last year eating habits before having been breast cancer diagnosed.
5. Physical activity study in the year prior to the diagnosis of breast cancer.
6. Anthropometric study: weight, size, waist circumference and body composition (% Fat mass,% Lean mass,% Body water).
7. Study of other risk factors of breast cancer: age, family history, reproductive history, medications consumed...
8. Biochemical study: biochemical variables of the last blood analysis performed on the volunteer in the hospital center.
9. Saliva collection to proceed with the genetic analysis.
10. Collection of stool sample to carry out the microbiota study.

ELIGIBILITY:
Inclusion Criteria:

* Older women than 18 years old
* Newly diagnosed patients with a breast tumor (Phase I, II or III). Being in one of the following cases:

  1. Patient who has not yet received any treatment and the committee has decided that as a first treatment will receive chemo or radiotherapy.
  2. Patient who has just undergone surgery and is waiting to start adjuvant treatment with chemo or radiotherapy.
* Sign the informed consent.

Exclusion Criteria:

* Patients with stage IV disease.
* Associated Eating Disorders.
* Patients with dementia, mental illness or decreased cognitive function.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a recent diagnosis of breast cancer
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dietary habits of a group of women with pre and post-surgical breast cancer | Six months
  Frequency of Consumption of food questionnaire referring. The frequency varies between one time per day and one time per month for every type of food during the last 6 months.
  to the last year of the volunteer's eating habits before being breast cancer diagnosed

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, Msc, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided